CLINICAL TRIAL: NCT01118780
Title: Duloxetine Versus Placebo in the Treatment of Elderly Patients With Generalized Anxiety Disorder
Brief Title: A Study of Duloxetine in Elderly Generalized Anxiety Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12866; F1J-MC-HMGF (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-05-05; First posted 2010-05-07 (Estimated); Results first posted 2013-09-02 (Estimated); Last update posted 2013-09-02 (Estimated); Status verified 2013-06

CONDITIONS: Generalized Anxiety Disorder
Keywords: GAD; Generalized Anxiety Disorder; Anxiety
MeSH Terms: conditions — Generalized Anxiety Disorder; Anxiety Disorders | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Duloxetine 30 milligrams (mg) -120 mg (Experimental)
  Interventions: Drug: Duloxetine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Duloxetine — Administered by mouth, daily for 10 weeks
  Other Names: Cymbalta; Duloxetine Hydrochloride; LY248686
  Arms: Duloxetine 30 milligrams (mg) -120 mg
Drug: Placebo — Administered by mouth, daily for 10 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to test the safety and efficacy of duloxetine versus placebo in elderly patients suffering from generalized anxiety disorder (GAD).

ELIGIBILITY:
Inclusion Criteria:

* Have GAD based on diagnostic criteria and not suffer from an adjustment disorder or anxiety disorder not otherwise specified. Symptoms of GAD should not be situational in nature.
* Have a Mini Mental State Examination (MMSE) score of at least 24 at screening.
* Have a Clinical Global Impressions of Severity (CGI-Severity) score of greater than or equal to 4 at screening and randomization.
* Have a Covi Anxiety Scale (CAS) score of greater than or equal to 9, no item in the Raskin Depression Scale (RDS) may be >3, and the CAS score must be greater than the RDS at screening.
* Have a Hospital Anxiety and Depression Scale (HADS) anxiety subscale score of greater than or equal to 10 at screening.
* Have a degree of understanding such that the participant can communicate intelligibly with the investigator and study coordinator.
* Are judged to be reliable to keep all appointments and able to swallow all required medication without opening or crushing.

Exclusion Criteria:

* Have any current and primary Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition-Text Revised (DSM-IV TR) Axis I diagnosis other than GAD, with the exception of comorbid social phobia or specific phobia.

  * major depressive disorder (MDD) within the past 6 months, or
  * panic disorder, posttraumatic stress disorder (PTSD), or an eating disorder within the past year, or
  * obsessive compulsive disorder (OCD), bipolar affective disorder, psychosis, factitious disorder, or somatoform disorders during their lifetime.
* The presence of an Axis II disorder, or history of antisocial behavior, or participants who, in the opinion of the investigator, are poor medical or psychiatric risks for study compliance.
* Have organic mental disorder or mental retardation diagnosis.
* Use of benzodiazepine within 14 days prior to randomization.
* Are judged clinically to be at serious risk of harm to self or others.
* Are currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an off-label use of an investigational drug or device, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
* Have previously completed or withdrawn from this study or any other study investigating duloxetine or have previously been treated with duloxetine within the past year or participants with a lack of response or intolerability to duloxetine (for any approved indication) at a clinically appropriate dose for a minimum of 4 weeks.
* Have a history of alcohol or any psychoactive substance abuse or dependence within the past 6 months.
* Excessively use caffeine, in the opinion of the investigator.
* Have a positive urine drug screen (UDS) for any substances of abuse at screening.
* Have a serious medical illness.
* Have any acute liver injury or severe cirrhosis.
* Have an abnormal thyroid-stimulating hormone (TSH) concentrations.
* Have initiated psychotherapy or changed intensity of psychotherapy or other non-drug therapies (such as acupuncture or hypnosis) within 6 weeks prior to enrollment or at any time during the study.
* Have taken any excluded medication within 7 days prior to randomization.
* Have been treated with a monoamine oxidase inhibitor (MAOI) or fluoxetine within 30 days of randomization or potentially need to use an MAOI during the study or within 5 days of discontinuation of study drug.
* Exhibit a lack of response of the current episode of GAD to 2 or more adequate trials of antidepressants, benzodiazepines, or other anxiolytics at a clinically appropriate dose for a minimum of 4 weeks.
* Have a history of severe allergies, hypersensitivity to duloxetine or to any of the inactive ingredients; multiple adverse drug reactions; transcranial magnetic stimulation (TMS); history of seizures; or history of psychosurgery or electroconvulsive therapy (ECT) within 12 months.
* Have discontinued hormone replacement therapy within the previous 3 months.
* Have uncontrolled narrow-angle glaucoma.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 291 (Actual)
Dates: Start 2010-10; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (25):
- United States (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prairie Village, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashua, New Hampshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toms River, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Staten Island, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Clinton, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bellevue, Washington
- Argentina (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rosario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santiago del Estero
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vienna, Austria
- Canada (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sydney, Nova Scotia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chatham, Ontario
- Germany (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hattingen
- Mexico (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aguascalientes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
- Poland (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chełmno
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tuszyn
- Puerto Rico (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bayamón
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ponce
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chesterfield, Chesterfield, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study had 3 periods: a screening period (3 to 30 days prior to randomization, no study drug administered), a treatment period (10 weeks), and a taper period (2 weeks). Participants who completed the treatment period were considered to have completed the study. Participant Flow and results, unless specified otherwise, are during treatment period.
Groups:
- Duloxetine: 30 to 120 milligrams (mg) administered orally, once daily for 10 weeks. Starting dose, 30-mg capsule, once daily for 2 weeks, with option to increase dose (30-mg increments) at Weeks 2, 4, and 7. If participant's Clinical Global Impression of Improvement (CGI-Improvement) Score was ≥3 (minimal improvement, no change, or worse) at Week 2, 4, or 7, the dose was required to be increased by 30 mg. At end of 10-week treatment period, participants had choice to enter 2-week taper period or begin active treatment (duloxetine or other).
  Optional taper period: Dosing was dependent on the participant's final dosage during the treatment period. Participants taking duloxetine 120 or 90 mg once daily received duloxetine 60 mg once daily for 1 week followed by 30 mg once daily for 1 week. Participants taking duloxetine 60 mg once daily received duloxetine 30 mg once daily for 1 week followed by placebo for 1 week. Participants taking duloxetine 30 mg once daily received placebo for 2 weeks.
- Placebo: A placebo capsule administered orally, once daily for 10 weeks. At the end of the 10-week treatment period, participants had choice to enter the 2-week taper period (placebo capsule administered orally, once daily for 2 weeks) or begin active treatment (duloxetine or other).
Period: Overall Study
Arm/Group | Duloxetine | Placebo
Started | 151 | 140
Completed | 115 | 105
Not Completed | 36 | 35
Not completed — Adverse Event | 15 | 15
Not completed — Death | 1 | 0
Not completed — Lack of Efficacy | 2 | 6
Not completed — Physician Decision | 2 | 0
Not completed — Protocol Violation | 3 | 6
Not completed — Withdrawal by Subject | 13 | 8

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Duloxetine | Placebo | Total
Number analyzed (Participants) | 151 | 140 | 291
Age Continuous [Mean (Standard Deviation); unit: years] | 71.43 (5.39) | 71.70 (5.04) | 71.56 (5.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114 | 112 | 226
  Male | 37 | 28 | 65
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 55 | 47 | 102
  Not Hispanic or Latino | 96 | 93 | 189
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 17 | 18 | 35
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 0 | 5
  White | 129 | 120 | 249
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  Argentina | 17 | 12 | 29
  Austria | 13 | 10 | 23
  Canada | 10 | 8 | 18
  Germany | 20 | 20 | 40
  Mexico | 21 | 21 | 42
  Poland | 27 | 29 | 56
  Puerto Rico | 7 | 5 | 12
  Spain | 9 | 9 | 18
  United Kingdom | 10 | 7 | 17
  United States | 17 | 19 | 36
Hamilton Anxiety Rating Scale (HAMA) Total Score [Mean (Standard Deviation); unit: units on a scale] — The Structured Interview Guide for the Hamilton Anxiety Rating Scale (SIGH-A) was used to collect HAMA data. The HAMA Total Score consisted of 14 items that assessed the severity of anxiety. Each item was scored using a 5-point scale (0=not present to 4=very severe). The HAMA Total Score could have ranged from 0 to 56 and higher scores indicated a greater degree of symptom severity.
  units on a scale | 24.62 (6.40) | 24.36 (7.11) | 24.49 (6.74)
Years Since Onset of Generalized Anxiety Disorder (GAD) [Mean (Standard Deviation); unit: years] — GAD was defined as excessive anxiety and worry, present more days than not, for at least 6 months, in accordance with the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition-Text Revised (DSM-IV TR). The excessive anxiety and worry must have been difficult to control and must have caused significant distress or impairment in normal functioning.
  years | 12.78 (16.40) | 11.83 (14.55) | 12.32 (15.52)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 10 in Hamilton Anxiety Rating Scale (HAMA) Total Score
Description: The Structured Interview Guide for the Hamilton Anxiety Rating Scale (SIGH-A) was used to collect HAMA data. The HAMA consisted of 14 items that assessed the severity of anxiety. Each item was scored using a 5-point scale (0=not present to 4=very severe). The HAMA Total Score could have ranged from 0 to 56 and higher scores indicated a greater degree of symptom severity. Least squares (LS) mean were calculated and analyzed using mixed-model repeated measures (MMRM) adjusted for treatment, pooled investigator, age category, visit, treatment-by-visit, baseline score, and baseline-by-visit.
Time Frame: Baseline, Week 10
Population: Randomized participants with a baseline and at least 1 post-baseline HAMA Total Score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 143 | 131
units on a scale | -15.86 (0.63) | -11.69 (0.67)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS mean difference = 4.17, 95% CI 2-sided [2.47 to 5.88], Standard Error of Mean 0.86 — LS mean difference was calculated by placebo minus duloxetine. Positive values indicated improvement over placebo

2. Secondary Outcome: Change From Baseline to Week 10 in Sheehan Disability Scale (SDS) Global Functional Impairment Score
Description: The SDS was a participant-rated questionnaire used to assess the effect of the participant's symptoms on work/school (Item 1), social life/leisure activities (Item 2), and family/home management (Item 3). Each item was rated on a visual analog scale (VAS) from 0 (not at all) to 10 (very severely). The SDS Global Functional Impairment Score (SDS Global Score) was the sum of the 3 items and could have ranged from 0 (unimpaired) to 30 (highly impaired). Higher values indicated a higher functional impairment in the participant's work/social/family life. Least squares (LS) mean were calculated and analyzed using mixed-model repeated measures (MMRM) adjusted for treatment, pooled investigator, age category, visit, treatment-by-visit, baseline score, and baseline-by-visit.
Time Frame: Baseline, Week 10
Population: Randomized participants with a baseline and at least 1 post-baseline SDS Global Functional Impairment Score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 140 | 131
units on a scale | -8.60 (0.60) | -5.37 (0.64)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS mean difference = 3.23, 95% CI 2-sided [1.61 to 4.85], Standard Error of Mean 0.82 — LS mean difference was calculated by placebo minus duloxetine. Positive values indicated improvement over placebo

3. Secondary Outcome: Change From Baseline to Week 10 in Hamilton Anxiety Rating Scale (HAMA) (Psychic Anxiety Factor Score, Somatic Anxiety Factor Score, and Individual Item Scores: Anxious Mood Item and Tension Item)
Description: The Structured Interview Guide for the Hamilton Anxiety Rating Scale (SIGH-A) was used to collect HAMA data. The HAMA consisted of 14 items that assessed the severity of anxiety. Each item was scored using a 5-point scale (0=not present to 4=very severe). The HAMA Psychic Anxiety Factor Score was the sum of Items 1 to 6 and Item 14 and could have ranged from 0 to 28. The HAMA Somatic Anxiety Factor Score was the sum of Items 7 to 13 and could have ranged from 0 to 28. The HAMA Anxious Mood Item Score was the score for Item 1 and the HAMA Tension Item Score was the score for Item 2. In each case, higher scores indicated a greater degree of symptom severity. Least squares (LS) mean were calculated and analyzed using mixed-model repeated measures (MMRM) adjusted for treatment, pooled investigator, age category, visit, treatment-by-visit, baseline score, and baseline-by-visit.
Time Frame: Baseline, Week 10
Population: Randomized participants with a baseline and at least 1 post-baseline HAMA factor or item score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 143 | 131
units on a scale
  HAMA Psychic Anxiety Factor Score (n=143, 131) | -8.59 (0.36) | -6.19 (0.38)
  HAMA Somatic Anxiety Factor Score (n=143, 131) | -7.33 (0.33) | -5.57 (0.35)
  HAMA Anxious Mood Item Score (n=142, 131) | -1.77 (0.08) | -1.24 (0.09)
  HAMA Tension Item Score (n=143, 131) | -1.48 (0.08) | -1.17 (0.09)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The p-value is for the change from baseline to Week 10 in the HAMA Psychic Anxiety Factor Score; LS mean difference = 2.40, 95% CI 2-sided [1.43 to 3.37], Standard Error of Mean 0.49 — LS mean difference was calculated by placebo minus duloxetine. Positive values indicated improvement over placebo
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The p-value is for the change from baseline to Week 10 in the HAMA Somatic Anxiety Factor Score; LS mean difference = 1.76, 95% CI 2-sided [0.87 to 2.65], Standard Error of Mean 0.45 — LS mean difference was calculated by placebo minus duloxetine. Positive values indicated improvement over placebo
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The p-value is for the change from baseline to Week 10 in the HAMA Anxious Mood Item Score; LS mean difference = 0.52, 95% CI 2-sided [0.30 to 0.74], Standard Error of Mean 0.11 — LS mean difference was calculated by placebo minus duloxetine. Positive values indicated improvement over placebo
Statistical Analysis 4: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.007, Mixed Models Analysis — The p-value is for the change from baseline to Week 10 in the HAMA Tension Item Score; LS mean difference = 0.31, 95% CI 2-sided [0.09 to 0.53], Standard Error of Mean 0.11 — LS mean difference was calculated by placebo minus duloxetine. Positive values indicated improvement over placebo

4. Secondary Outcome: Change From Baseline to Week 10 Endpoint in Hospital Anxiety Depression Scale (HADS) Subscale Scores
Description: HADS was a 14-item questionnaire with 2 subscales (anxiety and depression). Each item was rated on a 4-point scale (0 to 3) and higher scores indicated a greater dysfunction. The HADS Anxiety Subscale Score was the sum of the odd numbered items and scores could have ranged from 0 to 21. The HADS Depression Subscale Score was the sum of the even numbered items and scores could have ranged from 0 to 21. Higher scores indicated a greater dysfunction. Least squares (LS) mean were calculated and analyzed using mixed-model repeated measures (MMRM) adjusted for treatment, pooled investigator, age category, visit, treatment-by-visit, baseline score, and baseline-by-visit.
Time Frame: Baseline, Week 10
Population: Randomized participants with a baseline and at least 1 post-baseline HADS Subscale Score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 143 | 132
units on a scale
  HADS Anxiety Subscale | -7.81 (0.37) | -5.62 (0.39)
  HADS Depression Subscale | -3.29 (0.29) | -1.61 (0.31)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The p-value is for the change from baseline to Week 10 in the HADS Anxiety Subscale Score; LS mean difference = 2.19, 95% CI 2-sided [1.20 to 3.18], Standard Error of Mean 0.50 — LS mean difference was calculated by placebo minus duloxetine. Positive values indicated improvement over placebo
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The p-value is for the change from baseline to Week 10 in the HADS Depression Subscale Score; LS mean difference = 1.69, 95% CI 2-sided [0.89 to 2.49], Standard Error of Mean 0.41 — LS mean difference was calculated by placebo minus duloxetine. Positive values indicated improvement over placebo

5. Secondary Outcome: Clinical Global Impressions of Improvement Scale (CGI-Improvement) at Week 10
Description: CGI-Improvement measured the clinician's perception of the participant's improvement at the time of assessment compared with the start of treatment. Scores could have ranged from 1 (very much improved) to 7 (very much worse). Least squares (LS) mean were calculated and analyzed using mixed-model repeated measures (MMRM) adjusted for treatment, pooled investigator, age category, visit, treatment-by-visit.
Time Frame: Week 10
Population: Randomized participants with at least 1 post-baseline CGI-Improvement Score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 143 | 132
units on a scale | 2.10 (0.10) | 2.63 (0.10)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS mean difference = 0.53, 95% CI 2-sided [0.26 to 0.79], Standard Error of Mean 0.14 — LS mean difference was calculated by placebo minus duloxetine. Positive values indicated improvement over placebo

6. Secondary Outcome: Patient's Global Impressions of Improvement Scale (PGI-Improvement) at Week 10
Description: PGI-Improvement measured the participant's perception of his or her improvement at the time of assessment compared with the start of treatment. Scores could have ranged from 1 (very much better) to 7 (very much worse). Least squares (LS) mean were calculated and analyzed using mixed-model repeated measures (MMRM) adjusted for treatment, pooled investigator, age category, visit, treatment-by-visit.
Time Frame: Week 10
Population: Randomized participants with at least 1 post-baseline PGI-Improvement Score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 143 | 132
units on a scale | 2.35 (0.11) | 2.97 (0.12)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS mean difference = 0.62, 95% CI 2-sided [0.33 to 0.91], Standard Error of Mean 0.15 — LS mean difference was calculated by placebo minus duloxetine. Positive values indicated improvement over placebo

7. Secondary Outcome: Change From Baseline to Week 10 in Brief Pain Inventory-Modified Short Form (BPI-SF) Pain Severity and Interference Subscales
Description: The BPI-SF Pain Severity Subscale was a participant-rated questionnaire that measured the severity of pain. Severity scores could have ranged from 0 (no pain) to 10 (pain as bad as you can imagine) for questions assessing worst pain, least pain, and average pain in the past 24 hours, and pain right now. The BPI-SF Interference Subscale measured the interference of pain with the participant's ability to function. Interference scores could have ranged from 0 (does not interfere) to 10 (completely interferes) for questions assessing interference of pain in the past 24 hours for general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. Least squares (LS) means were calculated and analyzed using mixed-model repeated measures (MMRM) adjusted for treatment, pooled investigator, age category, visit, treatment-by-visit, baseline score, and baseline-by-visit.
Time Frame: Baseline, Week 10
Population: Randomized participants with a baseline and at least 1 post-baseline BPI-SF Pain Severity or Interference Subscale Score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 141 | 132
units on a scale
  Worst Pain (n=141, 132) | -1.44 (0.21) | -0.90 (0.22)
  Least Pain (n=141, 132) | -0.92 (0.17) | -0.50 (0.19)
  Average Pain (n=141, 132) | -1.10 (0.18) | -0.68 (0.19)
  Pain Right Now (n=141, 132) | -0.81 (0.18) | -0.59 (0.20)
  General Activity (n=140, 131) | -1.45 (0.23) | -0.92 (0.24)
  Mood (n=140, 131) | -1.59 (0.22) | -1.19 (0.23)
  Walking Ability (n=140, 131) | -0.91 (0.23) | -0.31 (0.24)
  Normal Work (n=139, 131) | -1.21 (0.23) | -0.83 (0.24)
  Relations With Other People (n=140, 131) | -0.96 (0.21) | -0.80 (0.22)
  Sleep (n=140, 131) | -1.58 (0.27) | -1.07 (0.28)
  Enjoyment of Life (n=140, 131) | -1.74 (0.23) | -1.24 (0.24)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.059, Mixed Models Analysis — The p-value is for the change from baseline to Week 10 in BPI-SF Worst Pain Score; LS mean difference = 0.55, 95% CI 2-sided [-0.02 to 1.11], Standard Error of Mean 0.29 — LS mean difference was calculated by placebo minus duloxetine. Positive values indicated improvement over placebo
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.079, Mixed Models Analysis — The p-value is for the change from baseline to Week 10 in BPI-SF Least Pain Score; LS mean difference = 0.42, 95% CI 2-sided [-0.05 to 0.89], Standard Error of Mean 0.24 — LS mean difference was calculated by placebo minus duloxetine. Positive values indicated improvement over placebo
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.089, Mixed Models Analysis — The p-value is for the change from baseline to Week 10 in BPI-SF Average Pain Score; LS mean difference = 0.42, 95% CI 2-sided [-0.06 to 0.91], Standard Error of Mean 0.25 — LS mean difference was calculated by placebo minus duloxetine. Positive values indicated improvement over placebo
Statistical Analysis 4: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.371, Mixed Models Analysis — The p-value is for the change from baseline to Week 10 in BPI-SF Pain Right Now Score; LS mean difference = 0.23, 95% CI 2-sided [-0.27 to 0.73], Standard Error of Mean 0.25 — LS mean difference was calculated by placebo minus duloxetine. Positive values indicated improvement over placebo
Statistical Analysis 5: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.066, Mixed Models Analysis — The p-value is for the change from baseline to Week 10 in BPI-SF General Activity Score; LS mean difference = 0.53, 95% CI 2-sided [-0.04 to 1.09], Standard Error of Mean 0.29 — LS mean difference was calculated by placebo minus duloxetine. Positive values indicated improvement over placebo
Statistical Analysis 6: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.140, Mixed Models Analysis — The p-value is for the change from baseline to Week 10 in BPI-SF Mood Score; LS mean difference = 0.41, 95% CI 2-sided [-0.13 to 0.95], Standard Error of Mean 0.27 — LS mean difference was calculated by placebo minus duloxetine. Positive values indicated improvement over placebo
Statistical Analysis 7: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.040, Mixed Models Analysis — The p-value is for the change from baseline to Week 10 in BPI-SF Walking Ability Score; LS mean difference = 0.60, 95% CI 2-sided [0.03 to 1.18], Standard Error of Mean 0.29 — LS mean difference was calculated by placebo minus duloxetine. Positive values indicated improvement over placebo
Statistical Analysis 8: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.187, Mixed Models Analysis — The p-value is for the change from baseline to Week 10 in BPI-SF Normal Work Score; LS mean difference = 0.38, 95% CI 2-sided [-0.19 to 0.94], Standard Error of Mean 0.29 — LS mean difference was calculated by placebo minus duloxetine. Positive values indicated improvement over placebo
Statistical Analysis 9: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.515, Mixed Models Analysis — The p-value is for the change from baseline to Week 10 in BPI-SF Relations With Other People Score; LS mean difference = 0.17, 95% CI 2-sided [-0.34 to 0.68], Standard Error of Mean 0.26 — LS mean difference was calculated by placebo minus duloxetine. Positive values indicated improvement over placebo
Statistical Analysis 10: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.141, Mixed Models Analysis — The p-value is for the change from baseline to Week 10 in BPI-SF Sleep Score; LS mean difference = 0.50, 95% CI 2-sided [-0.17 to 1.18], Standard Error of Mean 0.34 — LS mean difference was calculated by placebo minus duloxetine. Positive values indicated improvement over placebo
Statistical Analysis 11: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.088, Mixed Models Analysis — The p-value is for the change from baseline to Week 10 in BPI-SF Enjoyment of Life Score; LS mean difference = 0.50, 95% CI 2-sided [-0.07 to 1.07], Standard Error of Mean 0.29 — LS mean difference was calculated by placebo minus duloxetine. Positive values indicated improvement over placebo

8. Secondary Outcome: Change From Baseline to Week 10 in Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF) Total Score
Description: The Q-LES-Q-SF was a participant-rated questionnaire designed to assess the degree of enjoyment and satisfaction experienced during the past week. The questionnaire consisted of 16 items rated on a 5-point scale ranging from 1 (very poor) to 5 (very good). The total raw score was the sum of Items 1 to 14 and could have ranged from 14 to 70. Total raw scores were converted to, and expressed as, the percentage of the maximum possible score. Percent=100*(total raw score - 14)/56. Higher scores indicated higher levels of enjoyment/satisfaction. Least squares (LS) mean were calculated and analyzed using analysis of covariance (ANCOVA) adjusted for treatment, pooled investigator, age category, and baseline.
Time Frame: Baseline, Week 10
Population: Randomized participants with a baseline and at least 1 post-baseline Q-LES-Q-SF Total Score; Last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: percent of maximum possible score
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 134 | 125
percent of maximum possible score | 15.11 (1.45) | 9.35 (1.52)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.002, ANCOVA; LS mean difference = -5.76, 95% CI 2-sided [-9.4 to -2.1], Standard Error of Mean 1.87 — LS mean difference was calculated by placebo minus duloxetine. Negative values indicated improvement over placebo

9. Secondary Outcome: Number of Participants With Treatment-Emergent Suicide-Related Ideation and Behavior Based on the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS captured the occurrence, severity, and frequency of suicide-related thoughts and behaviors. Suicidal ideation: a "yes" answer to any 1 of 5 suicidal ideation questions: wish to be dead, and 4 different categories of active suicidal ideation. Suicidal behavior: a "yes" answer to any 1 of 5 suicidal behavior questions: preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide. Treatment-emergent was the worsening or new occurrence of suicidal behavior or ideation during treatment compared with baseline (Week 0).
Time Frame: Baseline through 10 weeks
Population: Randomized participants with a baseline and at least 1 post-baseline C-SSRS Score.
Measure: Number; unit: participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 144 | 133
participants
  Treatment-Emergent Suicidal Ideation | 3 | 5
  Treatment-Emergent Suicidal Behavior | 0 | 0

10. Secondary Outcome: Change From Baseline to Week 10 in Sheehan Disability Scale (SDS) Work/School, Social Life, and Family/Home Management Individual Impairment Scores
Description: The SDS was a participant-rated questionnaire used to assess the effect of the participant's symptoms on work/school (Item 1), social life/leisure activities (Item 2), and family/home management (Item 3). Each item was rated on a visual analog scale (VAS) from 0 (not at all) to 10 (very severely). Higher values indicated a higher functional impairment in the participant's work/social/family life. Least squares (LS) mean were calculated and analyzed using mixed-model repeated measures (MMRM) adjusted for treatment, pooled investigator, age category, visit, treatment-by-visit, baseline score, and baseline-by-visit.
Time Frame: Baseline, Week 10
Population: Randomized participants with a baseline and at least 1 post-baseline SDS Work/School, Social Life/Leisure Activities, or Family/Home Management Individual Impairment Scores.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 140 | 131
units on a scale
  Work/School (n=56, 51) | -2.21 (0.33) | -1.08 (0.40)
  Social Life/Leisure Activities (n=140, 131) | -2.84 (0.22) | -1.94 (0.23)
  Family/Home Management (n=140, 131) | -2.82 (0.22) | -1.61 (0.24)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.010, Mixed Models Analysis — The p-value is for the change from baseline to Week 10 in SDS for Work/School Impairment Score; LS mean difference = 1.13, 95% CI 2-sided [0.27 to 1.98], Standard Error of Mean 0.43 — LS mean difference was calculated by placebo minus duloxetine. Positive values indicated improvement over placebo
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis — The p-value is for the change from baseline to Week 10 in SDS for Social Life/Leisure Activities Impairment Score; LS mean difference = 0.90, 95% CI 2-sided [0.32 to 1.48], Standard Error of Mean 0.29 — LS mean difference was calculated by placebo minus duloxetine. Positive values indicated improvement over placebo
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The p-value is for the change from baseline to Week 10 in SDS for Family/Home Management Impairment Score; LS mean difference = 1.21, 95% CI 2-sided [0.61 to 1.81], Standard Error of Mean 0.30 — LS mean difference was calculated by placebo minus duloxetine. Positive values indicated improvement over placebo

11. Secondary Outcome: Percentage of Participants With Response or Remission at Week 10 (Response and Remission Rates)
Description: Response was a ≥50% improvement (reduction) in the Hamilton Anxiety Rating Scale (HAMA) Total Score at treatment period endpoint compared with baseline. Two definitions were used to determine remission: Definition 1 (HAMA Total Score ≤7 at endpoint) and Definition 2 (HAMA Total Score ≤10 at endpoint). The Structured Interview Guide for the Hamilton Anxiety Rating Scale (SIGH-A) was used to collect HAMA data. The HAMA consisted of 14 items that assessed the severity of anxiety. Each item was scored using a 5-point scale (0=not present to 4=very severe). The HAMA Total Score could have ranged from 0 to 56 and higher scores indicated a greater degree of symptom severity.
Time Frame: Baseline, Week 10
Population: Randomized participants with a baseline and 1 post-baseline HAMA Total Score; Last observation carried forward (LOCF).
Measure: Number; unit: percentage of participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 143 | 132
percentage of participants
  Response | 71.3 | 45.5
  Remission (HAMA Total Score ≤7) | 44.8 | 29.5
  Remission (HAMA Total Score ≤10) | 62.2 | 40.2
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — The p-value is for percentage of participants having HAMA response at Week 10 and was adjusted for pooled investigator
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — The p-value is for percentage of participants having remission (HAMA Total Score ≤7) at Week 10 and was adjusted for pooled investigator
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — The p-value is for percentage of participants having remission (HAMA Total Score ≤10) at Week 10 and was adjusted for pooled investigator

12. Secondary Outcome: Percentage of Participants With Functional Remission at Week 10 (Functional Remission Rate)
Description: Two definitions, using the Sheehan Disability Scale (SDS) Global Functional Impairment Score (SDS Global Score), were used to determine functional remission: Definition 1 (SDS Global Score ≤5 at endpoint) and Definition 2 (SDS Global Score ≤6 at endpoint). The SDS was a participant-rated questionnaire used to assess the effect of the participant's symptoms on work/school (Item 1), social life/leisure activities (Item 2), and family/home management (Item 3). Each item was rated on a visual analog scale (VAS) from 0 (not at all) to 10 (very severely). The SDS Global Score was the sum of the 3 items and could have ranged from 0 (unimpaired) to 30 (highly impaired). Higher values indicated a higher functional impairment in the participant's work/social/family life.
Time Frame: Week 10
Population: All randomized participants with at least 1 post-baseline SDS Global Score; Last observation carried forward (LOCF).
Measure: Number; unit: percentage of participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 151 | 140
percentage of participants
  Functional Remission (SDS Global Score ≤5) | 55.0 | 32.9
  Functional Remission (SDS Global Score ≤6) | 60.9 | 40.7
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — The p-value is for the percentage of participants having functional remission (SDS Global Score ≤5) at Week 10 and was adjusted for pooled investigator
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — The p-value is for the percentage of participants having functional remission (SDS Global Score ≤6) at Week 10 and was adjusted for pooled investigator

13. Secondary Outcome: Percentage of Participants With Sustained Improvement (Sustained Improvement Rate)
Description: Two definitions, using the Hamilton Anxiety Rating Scale (HAMA) Total Score at endpoint compared with baseline, were used to determine sustained improvement: Definition 1 [sustained improvement overall required a ≥30% improvement (reduction) in the HAMA Total Score at treatment period endpoint, at an earlier visit prior to endpoint, and at all visits in between] and Definition 2 (sustained improvement from Week 2 required a ≥30% reduction at treatment period endpoint, at Week 2, and at all visits in between). Both definitions required at least 2 post-baseline visits. The Structured Interview Guide for the Hamilton Anxiety Rating Scale (SIGH-A) was used to collect HAMA data. The HAMA consisted of 14 items that assessed the severity of anxiety. Each item was scored using a 5-point scale (0=not present to 4=very severe). The HAMA Total Score could have ranged from 0 to 56 and higher scores indicated a greater degree of symptom severity.
Time Frame: (Baseline through 10 weeks) and (Baseline, Week 2 through Week 10)
Population: Randomized participants who had baseline and the required number of post-baseline HAMA Total Scores.
Measure: Number; unit: percentage of participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 134 | 124
percentage of participants
  Sustained Improvement Overall (n=134, 124) | 74.6 | 55.6
  Sustained Improvement From Week 2 (n=134, 123) | 26.9 | 17.9
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel — The p-value is for the percentage of participants having HAMA sustained improvement overall and was adjusted for pooled investigator
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.038, Cochran-Mantel-Haenszel — The p-value is for the percentage of participants having HAMA sustained improvement from Week 2 and was adjusted for pooled investigator

14. Secondary Outcome: Adverse Events (AEs) Leading to Discontinuation From Study
Description: The number of participants who discontinued from the study due to an AE (serious or other AE) during the treatment period. A summary of serious and other AEs is located in the Reported Adverse Events module.
Time Frame: Baseline through 10 weeks
Population: All randomized participants.
Measure: Number; unit: participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 151 | 140
participants | 16 | 15

15. Secondary Outcome: Percentage of Participants Reporting Falling Down
Description: The percentage of participants who reported 1 or more falls at or before Week 10.
Time Frame: Baseline through 10 weeks
Population: Randomized participants with no falls recorded at Baseline and at least 1 post-baseline assessment for falls.
Measure: Number; unit: percentage of participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 113 | 114
percentage of participants | 6.2 | 3.5

16. Other Pre Specified Outcome: Number of Participants Experiencing a Treatment-Emergent Adverse Event (AE) During the Taper Period
Description: Treatment-emergent AEs were newly occurring AEs or a worsening of AEs during the taper period. A summary of serious AEs and other AEs during the treatment period (baseline through 10 weeks) is located in the Reported Adverse Events module.
Time Frame: 2 weeks during the taper period
Population: Randomized participants who entered the taper period.
Measure: Number; unit: participants
Groups:
- Duloxetine 30 mg Then Placebo: Participants, whose final dose during the treatment period was duloxetine 60 mg, were administered a 30-mg duloxetine capsule orally, once daily for 1 week followed by a placebo capsule orally, once daily for 1 week, during the 2-week taper period.
- Duloxetine 60 mg Then 30 mg: Participants, whose final dose during the treatment period was 90 mg or 120 mg duloxetine, were administered duloxetine 60 mg (two 30-mg duloxetine capsules) orally, once daily for 1 week followed by a 30-mg duloxetine capsule orally, once daily for 1 week, during the 2-week taper period.
- Placebo: Participants, whose final dose during the treatment period was either placebo or duloxetine 30 mg, were administered a placebo capsule orally, once daily for 2 weeks, during the 2-week taper period.
Arm/Group | Duloxetine 30 mg Then Placebo | Duloxetine 60 mg Then 30 mg | Placebo
Number analyzed (Participants) | 31 | 34 | 114
participants
  Any Serious AE | 0 | 0 | 0
  Non-Serious AE, Dizziness | 1 | 1 | 1
  Non-Serious AE, Fatigue | 0 | 1 | 2
  Non-Serious AE, Hyperhidrosis | 0 | 0 | 2
  Non-Serious AE, Nausea | 0 | 1 | 1
  Non-Serious AE, Tinnitus | 2 | 0 | 0
  Non-Serious AE, Constipation | 0 | 0 | 1
  Non-Serious AE, Cystitis | 0 | 0 | 1
  Non-Serious AE, Headache | 0 | 0 | 1
  Non-Serious AE, Musculoskeletal Chest Pain | 0 | 1 | 0
  Non-Serious AE, Nightmare | 0 | 1 | 0
  Non-Serious AE, Oropharyngeal Pain | 0 | 1 | 0
  Non-Serious AE, Pain | 0 | 0 | 1
  Non-Serious AE, Vertigo | 1 | 0 | 0

17. Secondary Outcome: Time to First Response
Description: The time (days) to first response, defined as a ≥50% improvement (reduction) from baseline in the Hamilton Anxiety Rating Scale (HAMA) Total Score. Participants who did not have a response were censored at the last treatment period visit. The Structured Interview Guide for the Hamilton Anxiety Rating Scale (SIGH-A) was used to collect HAMA data. The HAMA consisted of 14 items that assessed the severity of anxiety. Each item was scored using a 5-point scale (0=not present to 4=very severe). The HAMA Total Score could have ranged from 0 to 56 and higher scores indicated a greater degree of symptom severity.
Time Frame: Baseline through 10 weeks
Population: All randomized participants. The number of censored participants (n)=36 participants in the duloxetine treatment arm and n=60 participants in the placebo treatment arm.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 151 | 140
days | 50.00 [48.00 to 51.00] | 70.00 [50.00 to 72.00]
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.005, Log Rank — The p-value was adjusted for pooled investigator

18. Secondary Outcome: Time to First Remission
Description: The time (days) to first remission. Two definitions, using the Hamilton Anxiety Rating Scale (HAMA) Total Score, were used to determine remission: Definition 1 (HAMA Total Score ≤7 at endpoint) and Definition 2 (HAMA Total Score ≤10 at endpoint). Participants who did not have remission were censored at the last treatment period visit. The Structured Interview Guide for the Hamilton Anxiety Rating Scale (SIGH-A) was used to collect HAMA data. The HAMA consisted of 14 items that assessed the severity of anxiety. Each item was scored using a 5-point scale (0=not present to 4=very severe). The HAMA Total Score could have ranged from 0 to 56 and higher scores indicated a greater degree of symptom severity.
Time Frame: Baseline through 10 weeks
Population: All randomized participants (pts). The number of censored pts (n)=72 pts in the duloxetine treatment arm and n=92 pts in the placebo treatment arm for time to first remission (HAMA Total Score ≤7) and n=49 pts in the duloxetine treatment arm and n=71 pts in the placebo treatment arm for the time to first remission (HAMA Total Score ≤10).
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 151 | 140
days
  Remission (HAMA Total Score ≤7) | 71.00 [69.00 to 72.00] | NA [72.00 to NA] — The median and upper confidence interval was not calculable because an insufficient number of participants reached the event (HAMA Total Score ≤7).
  Remission (HAMA Total Score ≤10) | 51.00 [50.00 to 57.00] | 71.00 [70.00 to 75.00]
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Log Rank — The p-value is for the time to first remission (HAMA Total Score ≤10) and was adjusted for pooled investigator

19. Secondary Outcome: Time to Sustained Improvement Overall
Description: Time (days) to the earliest visit at which the Hamilton Anxiety Rating Scale (HAMA) Total Score was a ≥30% improvement (reduction) from baseline that was sustained through the last treatment period visit. Participants who did not meet sustained improvement criteria were censored at the last treatment period visit. The Structured Interview Guide for the Hamilton Anxiety Rating Scale (SIGH-A) was used to collect HAMA data. HAMA consisted of 14 items that assessed the severity of anxiety. Each item was scored using a 5-point scale (0=not present to 4=very severe). The HAMA Total Score could have ranged from 0 to 56 and higher scores indicated a greater degree of symptom severity.
Time Frame: Baseline through 10 weeks
Population: All randomized participants. The number of participants censored (n)=43 participants in the duloxetine treatment arm and n=63 participants in the placebo treatment arm.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 151 | 140
days | 30.00 [29.00 to 48.00] | 50.00 [30.00 to NA] — The upper 95% confidence interval was not calculable due to an insufficient number of participants reaching the event by 10 weeks.
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.001, Log Rank — The p-value was adjusted for pooled investigator

20. Secondary Outcome: Time to First Functional Remission
Description: Time (days) to first functional remission. Two definitions, using the Sheehan Disability Scale (SDS) Global Functional Impairment Score (SDS Global Score), were used to determine functional remission: Definition 1 (SDS Global Score ≤5 at endpoint) and Definition 2 (SDS Global Score ≤6 at endpoint). Participants, who did not have an SDS Global Score ≤5 or ≤6, were censored at the last treatment period visit. The SDS was a participant-rated questionnaire used to assess the effect of the participant's symptoms on work/school (Item 1), social life/leisure activities (Item 2), and family/home management (Item 3). Each item was rated on a visual analog scale (VAS) from 0 (not at all) to 10 (very severely). The SDS Global Score was the sum of the 3 items and could have ranged from 0 (unimpaired) to 30 (highly impaired). Higher values indicated a higher functional impairment in the participant's work/social/family life.
Time Frame: Baseline through 10 weeks
Population: All randomized participants (pts). Number of pts censored (n)=50 pts in duloxetine treatment arm and n=73 pts in placebo treatment arm for time to first functional remission (SDS Global Score ≤5) and n=37 pts in duloxetine treatment arm and n=60 pts in placebo treatment arm time to first functional remission (SDS Global Score ≤6).
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 151 | 140
days
  Functional Remission (SDS Global Score ≤5) | 50.00 [48.00 to 68.00] | 72.00 [71.00 to NA] — The upper 95% confidence interval was not calculable because an insufficient number of participants had functional remission (SDS Global Score ≤5) by endpoint.
  Functional Remission (SDS Global Score ≤6) | 31.00 [29.00 to 49.00] | 71.00 [50.00 to 73.00]
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.006, Log Rank — The p-value is for the time to first functional remission (SDS Global Functional Impairment Score ≤5) and was adjusted for pooled investigator
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.003, Log Rank — The p-value is for time to first functional remission (SDS Global Functional Impairment Score ≤6) and was adjusted for pooled investigator

21. Secondary Outcome: Time to First Improvement
Description: The time (days) to first improvement, defined as a Clinical Global Impression of Improvement (CGI-Improvement) Score ≤2. Participants who did not have a CGI-I Score ≤2 were censored at the last treatment period visit. CGI-Improvement measured the clinician's perception of the participant's improvement at the time of assessment compared with the start of treatment. Scores could have ranged from 1 (very much improved) to 7 (very much worse). A CGI-Improvement Score of ≤2 was much improved or very much improved.
Time Frame: Baseline through 10 weeks
Population: All randomized participants. The number of participants censored (n)=37 participants in the duloxetine treatment arm and n=58 participants in the placebo treatment arm.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 151 | 140
days | 31.00 [29.00 to 50.00] | 52.00 [49.00 to 71.00]
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Log Rank — The p-value was adjusted for pooled investigator

ADVERSE EVENTS:
Time Frame: Baseline through 10 weeks.
Description: Serious adverse events and other adverse events during the treatment period. Refer to the Other Pre-Specified Outcome Measure 21 for a summary of serious adverse events and other adverse events during the taper period.
Arm/Group | Duloxetine | Placebo
Serious Adverse Events (participants affected / at risk) | 3/151 | 0/140
Other Adverse Events (participants affected / at risk) | 89/151 | 71/140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine (N=151) | Placebo (N=140)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) — Event resulted in death
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine (N=151) | Placebo (N=140)
Vertigo (Ear and labyrinth disorders) | 5 (5) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 6 (6) | 4 (4)
Constipation (Gastrointestinal disorders) | 14 (14) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 7 (8) | 5 (5)
Dry mouth (Gastrointestinal disorders) | 11 (11) | 2 (2)
Nausea (Gastrointestinal disorders) | 17 (18) | 9 (9)
Nasopharyngitis (Infections and infestations) | 3 (3) | 10 (10)
Fall (Injury, poisoning and procedural complications) | 6 (9) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 6 (6) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (6)
Dizziness (Nervous system disorders) | 12 (13) | 10 (11)
Headache (Nervous system disorders) | 16 (18) | 9 (10)
Somnolence (Nervous system disorders) | 9 (9) | 3 (3)
Insomnia (Psychiatric disorders) | 2 (2) | 7 (7)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days